CLINICAL TRIAL: NCT04384289
Title: The Effects of Nurse Led Transitional Care Model on Elderly Patients Undergoing Open Heart Surgery: A Randomized Controlled Trial
Brief Title: Nurse Led Transitional Care Model in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AIBU-KDC-SC01
Record Dates: First submitted 2020-04-05; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Nursing Care; Quality of Life; Transitional Care
Keywords: Transitional Care Model; heart surgery; nursing care; autonomy; quality of life; elderly

STUDY DESIGN:
Intervention Model Description: Randomized controlled intervention study with a parallel group in a pretest-posttest design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ''Standard Care'' (No Intervention): ''Standard Care'' group were given standard care services.
- "Transitional Care Model" (Experimental): "Transitional Care Model" group were given care based on the Transitional Care Model until the post discharge 9th week starting from date of hospitalization.
  Interventions: Procedure: Nursing care based on the Transitonal Care Model

INTERVENTIONS:
Procedure: Nursing care based on the Transitonal Care Model — Nursing care carried out in collaboration with a multidisciplinary team in line with Transitonal Care Model for elderly patients who have undergone open heart surgery
  Arms: "Transitional Care Model"

SUMMARY:
To evaluate the effectiveness of Nurse Led Transitional Care Model (TCM) on the functional autonomy, quality of life and rehospitalization rates of elderly patients undergoing open heart surgery.

DETAILED DESCRIPTION:
Rate and number of successful cases in open heart surgery has been increasing due to the advances in medical technology and surgery. To improve patient convalescence results and reduce rate of post-discharge readmission to hospital and unplanned post-discharge rehospitalization, home-care and follow-up process of patients should be managed successfully.

A total of 66 elderly patients who agreed to participate in the study between November 2017 and December 2018 were randomly assigned to the intervention (n: 33) and control (n: 33) groups. Patients in intervention group were given care based on the TCM until the post discharge 9th week starting from date of hospitalization. Patients in control group were given standard care services. Functional autonomy and quality of life levels of patients were evaluated at admission to the clinic and at the post-discharge 9th week whereas their repeated admission rates to the clinic and re-hospitalization rates were evaluated at post discharge 2nd, 6th and 9th weeks and finally 6 months. The CONSORT checklist was used to check the procedure.

ELIGIBILITY:
Inclusion Criteria:

* be hospitalized for the first time and for elective open heart surgery;
* have no other surgical intervention other than an open heart surgery,
* have no psychological and mental disorders,
* have no major chronic problems such as kidney problems, neurological problems or cancer,
* be able to speak Turkish,
* be available to be communicated by phone,
* provide consent to participate in the study,
* live at a maximum distance of 50 km from the hospital (for easy access during post-discharge follow-up visits).

Exclusion Criteria:

* ask to leave the study,
* be exposed to a disease or trauma that may affect his/her functional autonomy during the study,
* die throughout the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline(up to 24 hours after the admission) in functional autonomy on the Functional Autonomy Measurement System (SMAF) at 9th week after discharge. | Baseline(up to 24 hours after the admission) and Week 9 after discharge
  The Functional Autonomy Measurement System (SMAF) is a validated, self reported instrument assessing 25 functions of the individual including daily life activities, communication and mental functions. Possible scores range from 0 to -87. A total score below -5 obtained by the elderly person indicates that the patient is at the risk of losing his/her functional autonomy. Change = ( Week 9 after discharge score -Baseline score)

SECONDARY OUTCOMES:
Change from Baseline(up to 24 hours after the admission) inquality of life on the SF-36 Quality of Life Scale at 9th week after discharge. | Baseline(up to 24 hours after the admission) and Week 9 after discharge
  The SF-36 Quality of Life Scale is a validated, self reported instrument consists of 36 items in total, assessing the health status in eight aspects namely; physical function (10 items), social function (2 items), role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items) and overall health items (5 items). Each part of the scale is evaluated differently and hence does not have a total score that can be calculated. Change = ( Week 9 after discharge score -Baseline score).

OTHER OUTCOMES:
Repeated admission and rehospitalization rates | Post discharge 2nd, 6th and 9th weeks and finally 6 months
  The rate of repeated post discharge referrals to hospital and rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: SERGÜL DUYGULU, Assoc. Prof, Study Director — the advisor of this doctoral thesis study
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Town Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naylor MD, Hirschman KB, Hanlon AL, Bowles KH, Bradway C, McCauley KM, Pauly MV. Effects of alternative interventions among hospitalized, cognitively impaired older adults. J Comp Eff Res. 2016 May;5(3):259-72. doi: 10.2217/cer-2015-0009. Epub 2016 May 5. PMID 27146416
- [Background] Naylor MD, Aiken LH, Kurtzman ET, Olds DM, Hirschman KB. The care span: The importance of transitional care in achieving health reform. Health Aff (Millwood). 2011 Apr;30(4):746-54. doi: 10.1377/hlthaff.2011.0041. PMID 21471497
- [Result] Zhang P, Xing FM, Li CZ, Wang FL, Zhang XL. Effects of a nurse-led transitional care programme on readmission, self-efficacy to implement health-promoting behaviours, functional status and life quality among Chinese patients with coronary artery disease: A randomised controlled trial. J Clin Nurs. 2018 Mar;27(5-6):969-979. doi: 10.1111/jocn.14064. Epub 2018 Jan 8. PMID 28880419
- [Result] Zhang P, Hu YD, Xing FM, Li CZ, Lan WF, Zhang XL. Effects of a nurse-led transitional care program on clinical outcomes, health-related knowledge, physical and mental health status among Chinese patients with coronary artery disease: A randomized controlled trial. Int J Nurs Stud. 2017 Sep;74:34-43. doi: 10.1016/j.ijnurstu.2017.04.004. Epub 2017 Apr 14. PMID 28601691
- [Result] Wong FK, Yeung SM. Effects of a 4-week transitional care programme for discharged stroke survivors in Hong Kong: a randomised controlled trial. Health Soc Care Community. 2015 Nov;23(6):619-31. doi: 10.1111/hsc.12177. Epub 2014 Dec 3. PMID 25470529
- [Result] Sawatzky JA, Christie S, Singal RK. Exploring outcomes of a nurse practitioner-managed cardiac surgery follow-up intervention: a randomized trial. J Adv Nurs. 2013 Sep;69(9):2076-87. doi: 10.1111/jan.12075. Epub 2013 Jan 14. PMID 23317314
- [Result] Naylor MD, Brooten DA, Campbell RL, Maislin G, McCauley KM, Schwartz JS. Transitional care of older adults hospitalized with heart failure: a randomized, controlled trial. J Am Geriatr Soc. 2004 May;52(5):675-84. doi: 10.1111/j.1532-5415.2004.52202.x. PMID 15086645
- [Result] Naylor MD, Feldman PH, Keating S, Koren MJ, Kurtzman ET, Maccoy MC, Krakauer R. Translating research into practice: transitional care for older adults. J Eval Clin Pract. 2009 Dec;15(6):1164-70. doi: 10.1111/j.1365-2753.2009.01308.x. PMID 20367721
- [Result] Naylor MD, Hirschman KB, Hanlon AL, Bowles KH, Bradway C, McCauley KM, Pauly MV. Comparison of evidence-based interventions on outcomes of hospitalized, cognitively impaired older adults. J Comp Eff Res. 2014 May;3(3):245-57. doi: 10.2217/cer.14.14. PMID 24969152
- [Result] Lie I, Danielsen SO, Tonnessen T, Solheim S, Leegaard M, Sandvik L, Wisloff T, Vangen J, Rosstad TH, Moons P. Determining the impact of 24/7 phone support on hospital readmissions after aortic valve replacement surgery (the AVRre study): study protocol for a randomised controlled trial. Trials. 2017 May 30;18(1):246. doi: 10.1186/s13063-017-1971-y. PMID 28693599
- [Derived] Coskun S, Duygulu S. The effects of Nurse Led Transitional Care Model on elderly patients undergoing open heart surgery: a randomized controlled trial. Eur J Cardiovasc Nurs. 2022 Jan 11;21(1):46-55. doi: 10.1093/eurjcn/zvab005. PMID 33821999
- See also: transitional care model protocol — https://www.nursing.upenn.edu/ncth/transitional-care-model/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT04384289/Prot_SAP_000.pdf